CLINICAL TRIAL: NCT00313677
Title: Clinical Trial Readiness for the Dystroglycanopathies
Status: Recruiting | Type: Observational
Sponsor: Katherine Mathews (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Katherine Mathews, Professor and Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 200510743; U54NS053672 (NIH)
Record Dates: First submitted 2006-04-10; First posted 2006-04-12 (Estimated); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Muscular Dystrophy
Keywords: muscular dystrophy; MD; fukutin-related protein gene; limb girdle; FKRP gene; congenital muscular dystrophy; childhood onset LGMD; adult onset LGMD; POMT1; POMT2; POMGnT1; LARGE; alpha dystroglycan; dystroglycanopathy; ISPD/CRPPA; DPM 1, 2 or 3; GMPPB; B3GNT1/B4GAT1; B3GALNT2; GTDC2/POMGnT2; TMEM5/RXYLT1; Fukutin; DAG1; POMK/SGK196; DOLK; TRAPPC11; GOSR2; INPP5K
MeSH Terms: conditions — Muscular Dystrophies; Muscular Dystrophy, Limb-Girdle, Type 2I; Walker-Warburg Syndrome; Muscular Dystrophy, Limb-Girdle, Type 2M

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — fibroblasts, whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to describe the early signs and symptoms of the dystroglycanopathies, and to gather information that will be required for future clinical trials.

DETAILED DESCRIPTION:
Muscular dystrophies are a diverse group of inherited disorders characterized by progressive muscle weakness and wasting. The disorders are caused by mutations, or changes, in genes. Genes are tiny pieces of inherited material (DNA) that direct the body to make certain kinds of proteins.

In this study, researchers will examine the clinical presentation of muscular dystrophy caused by abnormal glycosylation of alpha-dystroglycan. Patients with dystroglycanopathies could have mutations in any one of the more than 20 currently identified genes, or evidence of dystroglycanopathy in biopsied muscle tissue . Symptoms range from congenital muscular dystrophy that may involve the brain and eye, through an adult-onset limb girdle muscular dystrophy.

The study involves a clinical evaluation at the University of Iowa. The evaluation includes muscle strength and motor ability testing, lung function testing, quality of life and activity assessment, and a review of past medical history. Portions of this evaluation will be repeated on a yearly basis. Financial assistance is available for travel to Iowa City. Support is also available for genetic testing for people with a dystroglycanopathy diagnosis based on muscle or skin biopsy analysis.

Knowledge gained from this study will improve healthcare recommendations for people with dystroglycanopathies, and provide a baseline for further study, including potential treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Elevated CK (creatine kinase)
* Evidence of a dystroglycanopathy as determined by review of muscle pathology OR documented mutation in one of the known genes OR abnormal alpha-dystroglycan glycosylation in cultured fibroblasts
* Dystroglycanopathies are predicted to affect all racial and ethnic backgrounds, and all patients with dystroglycanopathies will be eligible for participation.
* Participants may be of any age, including children, and males and females will be recruited equally.
* Patients will have varying degrees of muscular weakness, but otherwise should be in relatively good health.

Exclusion Criteria:

* There are no exclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: neuromuscular care clinic
Sampling Method: Non-Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2006-04; Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
10 meter walk | through study completion, an average of 1 yea
  time to walk 10 meters without assistive device

SECONDARY OUTCOMES:
4 stair climb | through study completion, an average of 1 yea
  time to climb 4 stairs with or without use of rails

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Mathews, M.D., Principal Investigator — University of Iowa; Kevin Campbell, Ph.D., Study Director — Co-Investigator; Steven A. Moore, M.D. Ph.D., Study Director — Co-Investigator
Locations (1):
- University of Iowa, 200 Hawkins Drive, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crockett CD, Bertrand LA, Cooper CS, Rahhal RM, Liu K, Zimmerman MB, Moore SA, Mathews KD. Urologic and gastrointestinal symptoms in the dystroglycanopathies. Neurology. 2015 Feb 3;84(5):532-9. doi: 10.1212/WNL.0000000000001213. Epub 2015 Jan 7. PMID 25568299
- [Background] Mathews KD, Stephan CM, Laubenthal K, Winder TL, Michele DE, Moore SA, Campbell KP. Myoglobinuria and muscle pain are common in patients with limb-girdle muscular dystrophy 2I. Neurology. 2011 Jan 11;76(2):194-5. doi: 10.1212/WNL.0b013e3182061ad4. No abstract available. PMID 21220724
- [Background] Jensen BS, Willer T, Saade DN, Cox MO, Mozaffar T, Scavina M, Stefans VA, Winder TL, Campbell KP, Moore SA, Mathews KD. GMPPB-Associated Dystroglycanopathy: Emerging Common Variants with Phenotype Correlation. Hum Mutat. 2015 Dec;36(12):1159-63. doi: 10.1002/humu.22898. Epub 2015 Sep 23. PMID 26310427
- [Background] Brun BN, Willer T, Darbro BW, Gonorazky HD, Naumenko S, Dowling JJ, Campbell KP, Moore SA, Mathews KD. Uniparental disomy unveils a novel recessive mutation in POMT2. Neuromuscul Disord. 2018 Jul;28(7):592-596. doi: 10.1016/j.nmd.2018.04.003. Epub 2018 Apr 10. PMID 29759639
- [Background] Lee AJ, Jones KA, Butterfield RJ, Cox MO, Konersman CG, Grosmann C, Abdenur JE, Boyer M, Beson B, Wang C, Dowling JJ, Gibbons MA, Ballard A, Janas JS, Leshner RT, Donkervoort S, Bonnemann CG, Malicki DM, Weiss RB, Moore SA, Mathews KD. Clinical, genetic, and pathologic characterization of FKRP Mexican founder mutation c.1387A>G. Neurol Genet. 2019 Mar 1;5(2):e315. doi: 10.1212/NXG.0000000000000315. eCollection 2019 Apr. PMID 31041397
- [Background] Gonzalez-Perez P, Smith C, Sebetka WL, Gedlinske A, Perlman S, Mathews KD. Clinical and electrophysiological evaluation of myasthenic features in an alpha-dystroglycanopathy cohort (FKRP-predominant). Neuromuscul Disord. 2020 Mar;30(3):213-218. doi: 10.1016/j.nmd.2020.01.002. Epub 2020 Jan 25. PMID 32115343
- [Background] Hagedorn JL, Dunn TM, Bhattarai S, Stephan C, Mathews KD, Pfeifer W, Drack AV. Electroretinogram abnormalities in FKRP-related limb-girdle muscular dystrophy (LGMDR9). Doc Ophthalmol. 2023 Feb;146(1):7-16. doi: 10.1007/s10633-022-09909-4. Epub 2022 Nov 18. PMID 36399172
- [Background] Weiss RM, Kerber RE, Jones JK, Stephan CM, Trout CJ, Lindower PD, Staffey KS, Campbell KP, Mathews KD. Exercise-induced left ventricular systolic dysfunction in women heterozygous for dystrophinopathy. J Am Soc Echocardiogr. 2010 Aug;23(8):848-53. doi: 10.1016/j.echo.2010.05.007. Epub 2010 Jun 19. PMID 20646909
- [Background] Brun BN, Mockler SR, Laubscher KM, Stephan CM, Wallace AM, Collison JA, Zimmerman MB, Dobyns WB, Mathews KD. Comparison of brain MRI findings with language and motor function in the dystroglycanopathies. Neurology. 2017 Feb 14;88(7):623-629. doi: 10.1212/WNL.0000000000003609. Epub 2017 Jan 13. PMID 28087826
- [Background] Gedlinske AM, Stephan CM, Mockler SRH, Laubscher KM, Laubenthal KS, Crockett CD, Zimmerman MB, Mathews KD. Motor outcome measures in patients with FKRP mutations: A longitudinal follow-up. Neurology. 2020 Oct 13;95(15):e2131-e2139. doi: 10.1212/WNL.0000000000010604. Epub 2020 Aug 6. PMID 32764098
- [Background] Brun BN, Mockler SR, Laubscher KM, Stephan CM, Collison JA, Zimmerman MB, Mathews KD. Childhood Activity on Progression in Limb Girdle Muscular Dystrophy 2I. J Child Neurol. 2017 Feb;32(2):204-209. doi: 10.1177/0883073816677680. Epub 2016 Nov 22. PMID 27872178
- [Background] Libell EM, Bowdler NC, Stephan CM, Zimmerman MB, Gedlinske AM, Mathews KD. The outcomes and experience of pregnancy in limb girdle muscular dystrophy type R9. Muscle Nerve. 2021 Jun;63(6):812-817. doi: 10.1002/mus.27184. Epub 2021 Feb 10. PMID 33501999
- [Background] Libell EM, Richardson JA, Lutz KL, Ng BY, Mockler SRH, Laubscher KM, Stephan CM, Zimmerman BM, Edens ER, Reinking BE, Mathews KD. Cardiomyopathy in limb girdle muscular dystrophy R9, FKRP related. Muscle Nerve. 2020 Nov;62(5):626-632. doi: 10.1002/mus.27052. Epub 2020 Sep 10. PMID 32914449
- [Background] Coffey LN, Stephan CM, Zimmerman MB, Decker CK, Mathews KD. Diagnostic delay in patients with FKRP-related muscular dystrophy. Neuromuscul Disord. 2021 Dec;31(12):1235-1240. doi: 10.1016/j.nmd.2021.08.013. Epub 2021 Sep 6. PMID 34857438
- [Background] Reelfs AM, Stephan CM, Mockler SRH, Laubscher KM, Zimmerman MB, Mathews KD. Pain interference and fatigue in limb-girdle muscular dystrophy R9. Neuromuscul Disord. 2023 Jun;33(6):523-530. doi: 10.1016/j.nmd.2023.05.005. Epub 2023 May 19. PMID 37247532
- [Background] Carlson CR, McGaughey SD, Eskuri JM, Stephan CM, Zimmerman MB, Mathews KD. Illness-associated muscle weakness in dystroglycanopathies. Neurology. 2017 Dec 5;89(23):2374-2380. doi: 10.1212/WNL.0000000000004720. Epub 2017 Nov 3. PMID 29101272
- [Background] Reelfs AM, Stephan CM, Czech TM, Cox MO, Joseph S, Darbro BW, Moore SA, Campbell KP, Mathews KD. UDP-glucose dehydrogenase variants cause dystroglycanopathy. Ann Clin Transl Neurol. 2025 Jun;12(6):1302-1308. doi: 10.1002/acn3.70002. Epub 2025 Apr 17. PMID 40245099
- See also: U of Iowa Wellstone Muscular Dystrophy Specialized Research Center website — https://wellstone.medicine.uiowa.edu/